CLINICAL TRIAL: NCT01816763
Title: Effective Screening for Pain Study
Acronym: ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRE 12-030
Record Dates: First submitted 2013-03-11; First posted 2013-03-22 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Pain; Pain Management
Keywords: Health Care Quality, Access, and Evaluation; Primary Health Care; Medical Informatics
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- tablet based NRS pain one week, followed by nurse pain screen (Experimental): tablet-based patient self-report of the 'NRS pain one week'
  Interventions: Behavioral: NRS pain one week
- tablet based PEG, followed by nurse pain screen (Experimental): tablet-based enhanced pain screening with the PEG (pain intensity, emotional, and functional pain interference)
  Interventions: Behavioral: PEG
- DVPRS, followed by nurse pain screen (Experimental): Defense Veterans Pain Rating Scale on tablet followed by usual nursing staff documented pain screening with NRS pain now
  Interventions: Behavioral: DVPRS

INTERVENTIONS:
Behavioral: NRS pain one week — Eligible patients will be randomly assigned to complete a patient-reported 'NRS one week' on a tablet prior to making contact with a nursing staff vital signs screener.
  Arms: tablet based NRS pain one week, followed by nurse pain screen
Behavioral: PEG — Eligible patients will be assigned to complete a patient-reported enhanced pain screening with the PEG on a tablet prior to making contact with a nursing staff vital signs screener.
  Arms: tablet based PEG, followed by nurse pain screen
Behavioral: DVPRS — Eligible patients will be randomly assigned to complete a patient-reported 'DVPRS' on a tablet prior to making contact with a nursing staff vital signs screener.
  Arms: DVPRS, followed by nurse pain screen

SUMMARY:
In light of the importance of pain and widespread interest in patient-centeredness, the Department of Veterans Affairs (VA) has been emphasizing and successfully making pain and its management a routine feature of the health record and a focus of care. Awareness of pain and efforts to improve pain management rest on the VA's '5th Vital Sign' - a policy and practice of nursing staff routinely screening for 'pain now' at every health encounter using a 0-10 Numeric Rating Scale (NRS).

The team's previous research on VA's '5th Vital Sign' informs the specific design of this Effective Screening for Pain (ESP) study as well as the proposed research products.

Alternatives to the current pain screening approach may improve the sensitivity and specificity of screening for chronic pain. These alternatives include the nurse administered NRS with a one week look back period and a three item scale (PEG) incorporating intensity and emotional and physical interference. The PEG is very similar to the gold standard Brief Pain Inventory (BPI) from which it is derived, in its sensitivity, specificity, and sensitivity to change in detecting clinically important, functionally impairing pain.

The investigators plan to evaluate alternatives to the VA's current '5th Vital Sign' for pain screening, focusing on simple, feasible measures that can be used cross-sectionally for pain screening. In the setting of a primary care clinic, the investigators plan to cross-sectionally evaluate three arms - a tablet based DVPRS, a tablet computer-based NRS one week, and a tablet computer-based PEG. All arms will be compared with the nurse administered NRS.

DETAILED DESCRIPTION:
Background:

In light of the importance of pain and widespread interest in patient-centeredness, the Department of Veterans Affairs (VA) has been emphasizing and successfully making pain and its management a routine feature of the health record and a focus of care. Awareness of pain and efforts to improve pain management rest on the VA's '5th Vital Sign' - a policy and practice of nursing staff routinely screening for 'pain now' at every health encounter using a 0-10 Numeric Rating Scale (NRS).

The team's previous research on VA's '5th Vital Sign' informs the specific design of this Effective Screening for Pain (ESP) study as well as the proposed research products.

Alternatives to the current pain screening approach may improve the sensitivity and specificity of screening for chronic pain. These alternatives include the nurse administered NRS with a one week look back period and a three item scale (PEG) incorporating intensity and emotional and physical interference.

The investigators plan to evaluate alternatives to the VA's current '5th Vital Sign' for pain screening, focusing on simple, feasible measures that can be used cross-sectionally for pain screening. In the setting of a primary care clinic, the investigators plan to cross-sectionally evaluate three arms - a tablet based DVPRS, a tablet computer-based NRS one week, and a tablet computer-based PEG. All arms will be compared with the nurse administered pain now.

Objectives:

1) Qualitatively evaluate Veteran and multidisciplinary provider perspectives on pain screening and the use of the NRS vs. the PEG items, clinician-assessed vs. patient-reported pain 2a) Quantitatively assess, in a 3-arm randomized controlled primary care clinical team-based trial using tablets, the feasibility and completion rates, validity, and variability of pain information obtained comparing: Tablet-based vs. nurse-documented pain (e.g., 5th vital sign by tablet vs. clinician assessed) and the rate and severity of pain detected in tablet-based 'NRS one week' (Arm 1), tablet-based PEG (Arm 2), and DVPRS (Arm 3). Also pain, self-reported disability.

2b) Informed by Aims 1 and 2a, qualitatively evaluate provider perspectives on different pain reports to facilitate better pain management.

Methods:

The investigators are conducting a two phase mixed method study that will build on prior work to develop and test enhanced pain screening approaches for primary care and Patient Aligned Care Teams (PACTs). In the first (development) phase of the study, the investigators will conduct semi-structured qualitative interviews and focus groups with primary care clinicians, other primary care team members including non-provider staff, and primary care Veteran patients, to understand what patient-reported pain assessment data are most useful for clinical decision-making and how this pain information can best be integrated into primary care team processes, including the role of informatics to optimize primary care pain management and link pain screening to management. This will inform the development of the enhanced pain screening approaches used in the Aim 2 randomized controlled trial (RCT). The investigators will also submit the enhanced tablet-based pain screening approaches to usability testing by the University of California Office of Information Technology.

The second (testing) phase of the study will include a multisite RCT to test the final enhanced pain screening approaches (Arm 1 PEG; Arm 2 NRS 'pain now', Arm 3 DVPRS) compared with the NRS one week (all Arms), on patient and primary care clinician outcomes. The investigators will assess whether the approaches improve detection of pain-related impairment, and also the feasibility, acceptability, and provider and patient experience with enhanced screening.

Status:

The investigators have completed data collection, coding, and analyses for all Aims. They have presented some findings as conference posters and presentations and published several manuscripts.

Findings from Aim 1 were used to guide the development of a tablet-based pain screening survey that the investigators tested in Aim 2a as a randomized control trial. The investigators have have completed data collection, and are currently analyzing results.

ELIGIBILITY:
Inclusion Criteria:

* All Veterans are eligible to participate in the clinical trial when presenting for routine care in the primary care clinic at all sites (VA at Palo Alto, Minneapolis, and Portland).
* All are eligible who do not opt out of participation.
* All participants in the baseline tablet intervention will also be eligible for a one week follow up telephone interview - unless they are unable to complete a phone interview (see exclusions).
* For the qualitative Veteran component, all Veterans who can hear and respond in an interview are eligible.
* Providers/staff must be clinic and facility staff including administrative clerks, regular part time or full time employees in primary care who routinely participate in the care of Veterans who have painful conditions.

Exclusion Criteria:

* Veterans who meet either of the following exclusion criteria that may interfere with outcome assessment will be ineligible for the follow up telephone interview:

  * a) no working telephone (home, office, or mobile)
  * b) hearing impaired and unable to complete a phone survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl A. Lorenz, MD MSHS, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannitrapani KF, Ahluwalia SC, McCaa M, Pisciotta M, Dobscha S, Lorenz KA. Barriers to Using Nonpharmacologic Approaches and Reducing Opioid Use in Primary Care. Pain Med. 2018 Jul 1;19(7):1357-1364. doi: 10.1093/pm/pnx220. PMID 29059412
- [Background] Haverfield MC, Giannitrapani K, Timko C, Lorenz K. Patient-Centered Pain Management Communication from the Patient Perspective. J Gen Intern Med. 2018 Aug;33(8):1374-1380. doi: 10.1007/s11606-018-4490-y. Epub 2018 May 29. PMID 29845465
- [Background] Giannitrapani K, McCaa M, Haverfield M, Kerns RD, Timko C, Dobscha S, Lorenz K. Veteran Experiences Seeking Non-pharmacologic Approaches for Pain. Mil Med. 2018 Nov 1;183(11-12):e628-e634. doi: 10.1093/milmed/usy018. PMID 29590422
- [Background] Ahluwalia SC, Giannitrapani KF, Dobscha SK, Cromer R, Lorenz KA. "It Encourages Them to Complain": A Qualitative Study of the Unintended Consequences of Assessing Patient-Reported Pain. J Pain. 2018 May;19(5):562-568. doi: 10.1016/j.jpain.2017.12.270. Epub 2018 Feb 5. PMID 29421247
- [Background] Giannitrapani KF, Day RT, Azarfar A, Ahluwalia SC, Dobscha S, Lorenz KA. What Do Providers Want from a Pain Screening Measure Used in Daily Practice? Pain Med. 2019 Jan 1;20(1):68-76. doi: 10.1093/pm/pny135. PMID 30085285
- [Background] Giannitrapani KF, Glassman PA, Vang D, McKelvey JC, Thomas Day R, Dobscha SK, Lorenz KA. Expanding the role of clinical pharmacists on interdisciplinary primary care teams for chronic pain and opioid management. BMC Fam Pract. 2018 Jul 3;19(1):107. doi: 10.1186/s12875-018-0783-9. PMID 29970008
- [Result] Giannitrapani KF, Ahluwalia SC, Day RT, Pisciotta M, Dobscha S, Lorenz K. Challenges to teaming for pain in primary care. Healthc (Amst). 2018 Mar;6(1):23-27. doi: 10.1016/j.hjdsi.2017.06.006. Epub 2017 Jul 13. No abstract available. PMID 28711504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Research Assistants approached patients in the waiting rooms of primary care clinics (including women's health primary care clinics) at VA Palo Alto, Minneapolis, and Portland and queried them about their eligibility.
Groups:
- Tablet Based NRS Pain Now, Followed by Nurse Pain Screen: tablet-based patient self-report of the 'NRS pain now'
  NRS pain now: Eligible patients will be randomly assigned to complete a patient-reported 'NRS now' on a tablet prior to making contact with a nursing staff vital signs screener.
Period: Overall Study
Arm/Group | Tablet Based NRS Pain Now, Followed by Nurse Pain Screen | Tablet Based PEG, Followed by Nurse Pain Screen | DVPRS, Followed by Nurse Pain Screen
Started | 195 | 194 | 180
Completed | 191 | 179 | 169
Not Completed | 4 | 15 | 11
Not completed — The main reason for an incomplete survey | 4 | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tablet Based NRS Pain Now, Followed by Nurse Pain Screen | Tablet Based PEG, Followed by Nurse Pain Screen | DVPRS, Followed by Nurse Pain Screen | Total
Number analyzed (Participants) | 195 | 194 | 180 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (15.2) | 62.3 (15.7) | 59.9 (16.0) | 60 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 34 | 74
  Male | 169 | 180 | 146 | 495
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 1 | 11
  Not Hispanic or Latino | 174 | 172 | 165 | 511
  Unknown or Not Reported | 16 | 17 | 14 | 47

OUTCOME MEASURES:

1. Primary Outcome: Arm 1 (NRS Now), to Arm 2 (PEG), to Arm 3 (Defense Veterans Pain Rating Scale (e.g.,DVPRS) Differences Baseline Overall Pain Compared With Gold Standard Chronic Pain Grade Questionnaire Intensity Subscale Items (e.g., CPG Scale, Pain Intensity)
Description: pain (Numeric Rating Scale - NRS and PEG (full scale name) and Defense Veterans Pain Rating Scale - DVPRS measures) using overall pain derived from each of the three measures compared cross sectionally with the three pain intensity items and scale of the Chronic Pain Grade (CPG) questionnaire. The latter addresses pain 'now', average pain, and worst pain. All measures (NRS, PEG, DVPRS, and CPG) are scored from 0-10 where 0 equals no pain and 10 equals worst possible pain.). the NRS is a one item pain intensity measure, the PEG is a 3 item measure combining pain intensity, pain-related emotional and functional interference, and the DVPRS integrates pain intensity, pain interference, faces pain, and colormetric indicators on a 0-10 overall pain scale. The study used no subscales for the NRS, PEG, or DVPRS, and all values reported are total measure scores, computed as the average of items. We compare them to the pain intensity score of the CPG. Higher scores signify worse pain.
Time Frame: Baseline (e.g., time of clinic visit) measures were cross sectionally assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tablet Based NRS Pain Now: tablet-based patient self-report of the 'NRS pain now'
  NRS pain now: Eligible patients will be randomly assigned to complete a patient-reported 'NRS now' on a tablet prior to making contact with a nursing staff vital signs screener.
- Tablet Based PEG: tablet-based enhanced pain screening with the PEG (pain intensity, emotional, and functional pain interference)
  PEG: Eligible patients will be assigned to complete a patient-reported enhanced pain screening with the PEG on a tablet prior to making contact with a nursing staff vital signs screener.
- DVPRS: Defense Veterans Pain Rating Scale on tablet followed by usual nursing staff documented pain screening with NRS pain now
  DVPRS: Eligible patients will be randomly assigned to complete a patient-reported 'DVPRS' on a tablet prior to making contact with a nursing staff vital signs screener.
Arm/Group | Tablet Based NRS Pain Now | Tablet Based PEG | DVPRS
Number analyzed (Participants) | 195 | 194 | 180
units on a scale | 4.43 (2.81) | 4.32 (3) | 4.06 (2.75)

2. Secondary Outcome: Arm 1 (NRS Now), to Arm 2 (PEG), to Arm 3 (DVPRS) Differences in Number of Individuals Who Failed to Complete Pain Screen
Description: Number of persons who failed to complete (NRS and PEG and DVPRS measures). the measures vary in complexity as the NRS is one item, the PEG 3 items, and the DVPRS includes 10 items integrating color, faces pain, function, and intensity descriptions of pain. Measures are fully described in Outcome 1 description.
Time Frame: Baseline cross sectional comparison at the time of clinic visit
Measure: Number; unit: participants
Arm/Group | Tablet Based NRS Pain Now | Tablet Based PEG | DVPRS
Number analyzed (Participants) | 190 | 194 | 180
participants | 4 | 15 | 11

3. Secondary Outcome: Arm 1 (NRS Now), to Arm 2 (PEG), to Arm 3 (DVPRS) Number of Participants Who Rated Overall Functional Status Worse Relative to Peers Using the Gill Single Item Questionnaire
Description: descriptive analysis comparing overall pain rated by the three measures at Baseline (NRS, PEG, DVPRS), two of which include function (PEG and DVPRS), using the outcome of pre-specified single item of self-reported function compared to one's peers as validated by Gill et. al.. All pain outcome measures (NRS, PEG, DVPRS) are described fully in Outcome 1. Gill single item is not otherwise formally named. It is a 3 item scale querying "self rated activity level relative to peers" where the categories include "less active, about as active, and more active" and is scored as a categorical 0-2 rating where 2 is optimal and 0 is worst relative function.
Time Frame: Baseline cross-sectional comparison at time of clinic visit
Measure: Number; unit: participants
Groups:
- Tablet-based NRS Pain Now: tablet-based patient self-report of the 'NRS pain now'
- Tablet-based PEG: tablet-based enhanced pain screening with the PEG (pain intensity, emotional, and functional pain interference)
- DVPRS: Defense Veterans Pain Rating Scale on tablet followed by usual nursing staff documented pain screening with NRS pain now
Arm/Group | Tablet-based NRS Pain Now | Tablet-based PEG | DVPRS
Number analyzed (Participants) | 109 | 122 | 101
participants | 50 | 60 | 48

ADVERSE EVENTS:
Time Frame: During baseline data collection for each participant. There was no study observation period or followup because the intervention was a screening tool administered as part of the baseline interview.
Description: The only study intervention was administering a tablet based survey, and events were only monitored during baseline data collection for each participant. There was no study observation period or followup because the intervention was a screening tool administered as part of the Baseline interview.No adverse events occurred.
Arm/Group | Tablet Based NRS Pain Now, Followed by Nurse Pain Screen | Tablet Based PEG, Followed by Nurse Pain Screen | DVPRS, Followed by Nurse Pain Screen
All-Cause Mortality (participants affected / at risk) | 0/195 | 0/194 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/195 | 0/194 | 0/180
Other Adverse Events (participants affected / at risk) | 0/195 | 0/194 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT01816763/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT01816763/SAP_001.pdf